CLINICAL TRIAL: NCT04963595
Title: Phase II Study of Pyrotinib and Vinorelbine Tartrate Capsules With or Without Inetetamab for First Line Treatment in Patients With Trastuzumab-resistant HER2-positive Advanced Breast Cancer
Brief Title: Pyrotinib and Vinorelbine Tartrate Capsules With or Without Inetetamab for First Line Treatment in Patients With Trastuzumab-resistant HER2-positive Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhiyong Yu (Other)
Responsible Party: Sponsor-Investigator, Zhiyong Yu, Chief of breast department, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ShandongCHI-20
Record Dates: First submitted 2021-07-11; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Vinorelbine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyrotinib and Vinorelbine with Inetetamab (Experimental)
  Interventions: Drug: Pyrotinib; Drug: Vinorelbine; Drug: Inetetamab
- Pyrotinib and Vinorelbine without Inetetamab (Experimental)
  Interventions: Drug: Pyrotinib; Drug: Vinorelbine

INTERVENTIONS:
Drug: Pyrotinib — 400 mg once daily
Drug: Vinorelbine — Initial dose 70 mg/m2 on days 1 and 8 (capsules) If well tolerated, subsequently 90 mg/m2 on days 1 and 8. Capsules on day 1 to be taken at the hospital, and on day 8 at home.
Drug: Inetetamab — 8mg/kg iv day 1 followed by 6mg/kg iv day 1, cycled every 21 days
  Arms: Pyrotinib and Vinorelbine with Inetetamab

SUMMARY:
Trastuzumab resistance, which is a common therapeutic challenge in HER2 positive metastatic breast cancer, is not fully understood. Pyrotinib is an oral tyrosine kinase inhibitor targeting EGFR, HER-2 and HER-4 receptors. More general inhibition of ErbB family with pyrotinib could provide additional benefit. Inetetamab could bind to HER2 extracellular domain (ECD) with high affinity and inhibit proliferation of multiple HER2-overexpressing cancer cell lines as a single agent or in combination with trastuzumab. This study is designed to evaluate the efficacy and safety of pyrotinib and vinorelbine tartrate capsulesin with or without Inetetamab for first line treatment in patients with HER2 positive metastatic breast cancer who had early failure on or after trastuzumab treatment.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed invasive breast cancer HER2 status must be prospectively, centrally tested and be HER2-positive based on central laboratory assay results Prior treatment for breast cancer in the adjuvant, unresectable, locally advanced, or metastatic setting must include both a taxane, alone or in combination with another agent, and trastuzumab, alone or in combination with another agent. Patients who have previously used pertuzumab will be allowed.

Documented progression (which occur during or after most recent treatment or within 6 months after completing of adjuvant therapy) of incurable, unresectable, locally advanced or metastatic breast cancer, defined by the investigator Measurable and/or nonmeasurable disease; participants with central nervous system-only disease are excluded Cardiac ejection fraction greater than or equal to (>/=) 50 percent (%) by either echocardiogram or multi-gated acquisition scan Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

History of treatment with pyrotinib Prior treatment with lapatinib or neratinib History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma History of receiving any anti-cancer drug/biologic or investigational treatment within 28 days prior to randomization except hormone therapy Recovery of treatment-related toxicity consistent with other eligibility criteria History of radiation therapy within 28 days of randomization Brain metastases that are untreated, symptomatic, or require therapy to control symptoms, as well as any history of radiation, surgery, or other therapy, including steroids, to control symptoms from brain metastases within 2 months (60 days) of randomization History of symptomatic congestive heart failure or serious cardiac arrhythmia requiring treatment History of myocardial infarction or unstable angina Current severe, uncontrolled systemic disease (for example, clinically significant cardiovascular, pulmonary, or metabolic disease) Pregnancy or lactation Current known active infection with human immunodeficiency virus (HIV) or hepatitis C virus Presence of conditions that could affect gastrointestinal absorption: Malabsorption syndrome, resection of the small bowel or stomach, and ulcerative colitis

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
Objective Response Rate | 3 years
  from enrollment to progression or death (for any reason), assessed up to 3 years